CLINICAL TRIAL: NCT00946725
Title: A Comparative Bioavailability Study of Atenolol Tablets, 100 mg
Brief Title: To Demonstrate the Relative Bioavailability of Atenolol Tablets, 100 mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Eric Mittleberg, Ph.D, VP of Product Development, Sandoz Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 11627
Record Dates: First submitted 2009-07-24; First posted 2009-07-27 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2009-07

CONDITIONS: Angina; Hypertension
Keywords: Angina (Chest Pain); Hypertension
MeSH Terms: conditions — Angina Pectoris; Hypertension; Chest Pain | interventions — Atenolol

ARMS (2):
- 1 (Experimental): Atenolol 100 mg Tablets (Geneva Pharmaceutical, Inc.)
  Interventions: Drug: Atenolol 100 mg Tablets (Geneva Pharmaceutical, Inc.)
- 2 (Active Comparator): Atenolol (Tenormin) 100 mg Tablets Zeneca (Astra Zeneca Pharmaceutical)
  Interventions: Drug: Atenolol (Tenormin) 100 mg Tablets Zeneca (Astra Zeneca Pharmaceutical)

INTERVENTIONS:
Drug: Atenolol (Tenormin) 100 mg Tablets Zeneca (Astra Zeneca Pharmaceutical)
  Arms: 2
Drug: Atenolol 100 mg Tablets (Geneva Pharmaceutical, Inc.)
  Arms: 1

SUMMARY:
To demonstrate the relative bioavailability of atenolol tablets, 100 mg.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal finding on physical exam, medical history, or clinical laboratory results on screening.

Exclusion Criteria:

* Positive test results for HIV or hepatitis B or C.
* Treatment for drug or alcohol dependence.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2000-11; Primary Completion 2000-11 (Actual); Study Completion 2000-11 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on AUC and Cmax | 20 days

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Goldwater, M.D., Principal Investigator — PharmaKinetics Laboratories Inc.